CLINICAL TRIAL: NCT01128439
Title: A Postmarketing Observational Study Estimating The Impact Of Prevnar 13 (Trade Mark) (13vpnc) On Invasive Pneumococcal Disease Caused By Vaccine Serotypes Of Streptococcus Pneumoniae After Introduction Into Routine Pediatric Use
Brief Title: Study Estimating the Impact of Prevnar 13™ (13vPnC) on Invasive Pneumococcal Disease
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Kaiser Permanente (Other)
Responsible Party: Sponsor
Other Study IDs: 6096A1-4005; B1851042 (Other: Alias Study Number)
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2018-12-04 (Actual); Status verified 2018-11

CONDITIONS: Invasive Pneumococcal Disease
Keywords: Pneumococcal conjugate vaccine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study will estimate the incidence of invasive pneumococcal disease in members of the Northern Kaiser Permanente healthcare system during each of the 5 following introduction of Prevnar 13.

DETAILED DESCRIPTION:
No sampling as no subjects are enrolled

ELIGIBILITY:
Inclusion Criteria:

* Documented invasive pneumococcal disease (IPD), defined as recovery of an isolate of S pneumoniae from a normally sterile site in a member of the surveillance population.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Incidence of IPD in the NCKP healthcare system in children 6 weeks through 5 years of age (prior to the sixth birthday) during each of the 5 years following introduction of Prevnar 13. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Kaiser Permanente Vaccine Study Center, Oakland, California, United States

REFERENCES:
- [Derived] Baxter R, Aukes L, Pelton SI, Yee A, Klein NP, Gruber WC, Scott DA, Center KJ. Impact of the 13-Valent Pneumococcal Conjugate Vaccine on Invasive Pneumococcal Disease After Introduction Into Routine Pediatric Use. J Pediatric Infect Dis Soc. 2021 Mar 26;10(2):141-150. doi: 10.1093/jpids/piaa035. PMID 32415771